CLINICAL TRIAL: NCT01244698
Title: Postoperative Antibiotic Requirements Following Immediate Breast Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Principal Investigator, Duc T Bui, MD, Associate Professor of Surgery, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160583-3
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Bacterial Infection; Anti-infective Agents; Breast Implantation
Keywords: Surgical Site Infection, Breast Reconstruction, Antibiotics
MeSH Terms: conditions — Bacterial Infections; Surgical Wound Infection | interventions — Clindamycin; Cefadroxil; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics until Drain Removal (Other): All patients will receive 24 hours of IV Cefazolin, as is universal practice for clean breast surgery. The control group will receive oral outpatient Cefadroxil until the final drain is removed. In case of significant penicillin allergy (defined as a history of urticaria or anaphylaxis associated with penicillin) patients will receive Clindamycin.
  Interventions: Drug: Cefadroxil until drain removal
- Early discontinuation of antibiotics (Experimental): All patients will receive 24 hours of IV Cefazolin, as is universal practice for clean breast surgery. The interventional group will then discontinue antibiotics.
  Interventions: Drug: Cefadroxil discontinued early

INTERVENTIONS:
Drug: Cefadroxil discontinued early — All patients will receive 24 hours of IV Cefazolin (1g IV every 8 hr), as is universal practice for clean breast surgery. The interventional group will then discontinue antibiotics. Clindamycin IV 600mg every 6 hours for 24 hours will be used in penicillin allergic patients.
  Other Names: Clindamycin; Cleocin; Duricef; Ancef; Cefazolin
  Arms: Early discontinuation of antibiotics
Drug: Cefadroxil until drain removal — All patients will receive 24 hours of IV Cefazolin, as is universal practice for clean breast surgery. The control group will receive oral outpatient Cefadroxil (500mg 2 times a day) until the final drain is removed. This is the normal postoperative regimen. In case of significant penicillin allergy (defined as a history of urticaria or anaphylaxis associated with penicillin) patients will receive Clindamycin 600mg IV every 6 hours for 24 hours followed by clindamycin 300mg IV every 6 hours.
  Other Names: Duricef; Cefazolin; Ancef; Clindamycin; Cleocin
  Arms: Antibiotics until Drain Removal

SUMMARY:
Antibiotics are used routinely in postoperative tissue expander based breast reconstruction (TE) and autologous flap (AF) breast reconstruction procedures. Closed suction drains are also used routinely in immediate breast reconstruction to prevent fluid accumulation and seroma formation at the surgical sites. Antibiotics are most often prescribed as a precaution since drains can be a source for infection by creating open channels to outside contaminants. Plastic surgery patients without closed suction drainage devices are usually not placed on prolonged postoperative antibiotics. Current preoperative surgical antibiotic prophylaxis is recommended for up to 24 hours only. These recommendations do not take into account the increased risk of indwelling closed suction drains. A recent survey of plastic surgeons, conducted by SBUMC investigators, (IRB# 129415) found that Plastic Surgeons are divided as to extended outpatient administration following TE breast reconstruction.

The study plans to prospectively enroll patients who will undergo immediate breast reconstruction with TE or AF based breast reconstruction. Using the above data and the current protocol, the investigators will investigate the optimal antibiotic discontinuation period for these patients. The investigators hypothesize that the use of 24-hour perioperative antibiotics in TE or AF based immediate breast reconstruction with closed suction drainage, does not result in an increased infection rate compared to prolonged postoperative antibiotic administration.

DETAILED DESCRIPTION:
Background:

Antibiotics are used routinely in postoperative tissue expander based breast reconstruction (TE) and autologous flap (AF) breast reconstruction procedures. Closed suction drains are also used routinely in immediate breast reconstruction to prevent fluid accumulation and seroma formation at the surgical sites. Antibiotics are most often prescribed as a precaution because drains may serve as an open channel to outside contaminants. Plastic surgery patients without closed suction drainage devices are usually not placed on prolonged postoperative antibiotics. Current preoperative surgical antibiotic prophylaxis is recommended for up to 24 hours only. These recommendations do not take into account the increased risk of indwelling closed suction drains.

Current plastic surgery literature does not provide recommendations or consensus for antibiotic discontinuation following immediate breast reconstruction. A recent survey conducted of 650 plastic surgeons showed that 98% of respondents give preoperative antibiotics, while 91% provide antibiotics for up to 24 hours. Additionally, 71% of respondents prescribe postoperative outpatient antibiotics. There was a divide of when to discontinue antibiotics among plastic surgeons who gave them postoperatively. 46% preferred to continue antibiotics until drain removal, while 52% preferred a specific postoperative day, most commonly day 5 or 7.

In the same survey, the majority (97%) of surgeons use IV Cefazolin as the choice for preoperative prophylaxis and oral Cephalexin (75.4%) and Cefadroxil (14.3%) for outpatient antibiotics. Currently at Stony Brook University Medical Center, patients normally receive 24 hours of IV Cefazolin, followed by postoperative antibiotic prescription for Cefadroxil. Antibiotics are discontinued when the final drain is removed.

The study plans to prospectively enroll patients who will undergo immediate breast reconstruction with TE or AF based breast reconstruction. Using the above data and the current protocol, the investigators will investigate the optimal antibiotic discontinuation period for these patients. The investigators will randomize these patients into two groups. One group will receive the current antibiotic regimen of 24 hours of IV Cefazolin, followed by outpatient Cefadroxil. Antibiotics will be discontinued for this group once the final drain is removed. The other group will only receive 24 hours of IV Cefazolin without any additional outpatient antibiotics, as is recommended for elective clean surgeries. In patients with penicillin allergies or sensitivity, clindamycin, IV and oral is used. The same randomization will apply in these patients.

Rationale for early discontinuation of postoperative antibiotics:

Studies have associated prolonged antimicrobial prophylaxis with development of resistant bacterial strains following surgical procedures. No evidence has been reported supporting practices of continuing antibiotics until drains are removed. A single dose of preoperative IV antibiotics has been suggested to be sufficient prophylaxis for most breast surgery patients discharged home with drains.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Stony Brook University Medical Center Plastic Surgery clinic for immediate breast reconstruction using a tissue expander.
* Age 18 years or older

Exclusion Criteria

* Delayed or revision implant reconstruction
* Refusal or inability to consent
* Contraindications to surgery as determined by attending physician
* Contraindications to both penicillin/cephalosporin and clindamycin antibiotics (significant allergies)
* Patients with serious existing systemic infection, defined as 2 or more of the following:

Peripheral body temperature >38 degrees Celsius CRP >5g/L Leukocytes > 12,000/microliter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Surgical Site infection | 365 days after the procedure
  One or more of the following:
  1. Purulent drainage, with or without laboratory confirmation, from the superficial incision.
  2. Organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision.
  3. At least one of the following signs or symptoms of infection: pain or tenderness, localized swelling, redness, or heat and superficial incision is deliberately opened by surgeon, unless incision is culture-negative.
  4. Diagnosis of superficial incisional SSI by the surgeon or attending physician.

SECONDARY OUTCOMES:
Antibiotic Sensitivity | From administration of the antibiotic until discontinuation
  Assessed by documentation of an allergic or adverse sensitivity reaction including, but not limited to urticaria, itching, rash, anaphylaxis
Clostridium Difficile Colitis | up to 365 days postoperatively
  C. Difficile colitis will be assessed by documented positive c. difficile toxin assay.
Antibiotic Resistance | 1 year postoperatively
  Local wound infections will be cultured and sent for identification and susceptibility. Alternatively, pathological fluid collections will be aspirated and fluid will be sent for culture and susceptibility. Resistant strains will be documented and treated with alternative antibiotics.
Patient compliance | while antibiotics are being administered postoperatively
  patients will be asked to bring antibiotics to clinic for counting to assess compliance.
Cost | while antibiotics are being administered postoperatively
  Cost will be assessed by multiplying the duration of outpatient postoperative antibiotics by the cost for self-pay prescriptions.

CONTACTS AND LOCATIONS:
Overall Officials: Duc T Bui, MD, Principal Investigator — Stony Brook University Medical Center; Brett T Phillips, MD, Study Director — Stony Brook University Medical Center; Duc T Bui, MD, Study Chair — Stony Brook University Medical Center
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States

REFERENCES:
- [Derived] Phillips BT, Fourman MS, Bishawi M, Zegers M, O'Hea BJ, Ganz JC, Huston TL, Dagum AB, Khan SU, Bui DT. Are Prophylactic Postoperative Antibiotics Necessary for Immediate Breast Reconstruction? Results of a Prospective Randomized Clinical Trial. J Am Coll Surg. 2016 Jun;222(6):1116-24. doi: 10.1016/j.jamcollsurg.2016.02.018. Epub 2016 Mar 4. PMID 27106640